CLINICAL TRIAL: NCT00391430
Title: Cognitive Behavioral Therapy vs. Sertraline in the Treatment of Post Traumatic Stress Disorder
Brief Title: Cognitive Behavioral Therapy Versus Sertraline in the Treatment of Post-Traumatic Stress Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty enrolling subjects
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: P50MH058911 (NIH); P50MH058911 (NIH); DATR A3-NSC
Record Dates: First submitted 2006-10-20; First posted 2006-10-24 (Estimated); Results first posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-06

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; Trauma; Sexual Abuse; Sexual Assault
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Sertraline; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Control (No Intervention): Participants assigned to the control condition will receive no treatment
- Sertraline (Active Comparator): Participants will receive treatment with sertraline
  Interventions: Drug: Sertraline
- CBT (Active Comparator): Participants will receive cognitive behavioral therapy
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)

INTERVENTIONS:
Drug: Sertraline — Dosage: up to 100 mg/day; Frequency: once per day; Duration: 12 weeks
  Arms: Sertraline
Behavioral: Cognitive behavioral therapy (CBT) — CBT consists of sixteen 1-hour sessions during a period of 12 weeks.
  Arms: CBT

SUMMARY:
This study will evaluate which parts of the brain are affected by treatment with behavioral therapy versus medication therapy in people with post-traumatic stress disorder.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is an anxiety disorder that can develop after exposure to a traumatic event. PTSD symptoms may include emotional numbness, loss of interest in activities that were once enjoyable, irritability, and sleep problems. Medication therapy, behavioral therapy, and a combination of both therapies are among the available treatment options for people with PTSD. Cognitive behavioral therapy (CBT), a type of talking therapy that has been shown to be effective in treating PTSD, teaches patients how to alter their thinking to, in turn, improve how they feel. A selective serotonin reuptake inhibitor (SSRI) is a type of medication that has also been effective in treating PTSD. Information about the comparative physiological effects of each of these treatments on people with PTSD is needed. This study will evaluate which parts of the brain are affected by CBT treatment versus SSRI treatment in people with PTSD.

Participants with and without PTSD will be enrolled in this 12-week, open label study. Following a screening visit to determine eligibility, participants with PTSD will be offered a choice of either CBT or SSRI treatment. Those participants who choose CBT will attend 16 therapy sessions. The first phase of therapy will focus on the development of emotional and interpersonal regulation skills. The second phase will use a modified form of prolonged exposure therapy, which has been effective in reducing symptoms of PTSD. Participants who elect to receive medication will take sertraline, an SSRI that has been safe and effective in treating PTSD. These participants will attend 12 treatment sessions. Pre- and post-treatment fear response will be assessed in all participants using fMRI scans to measure brain responses and using saliva samples to test cortisol levels. All participants will also self-administer saliva samples at various points during the 3 days prior to fMRI scanning. Other outcomes will be assessed throughout the study using questionnaires.

For information on a related study, please follow this link:

http://clinicaltrials.gov/show/NCT00648375

ELIGIBILITY:
Inclusion Criteria:

For people with PTSD:

* Meets DSM-IV criteria for PTSD
* Medically healthy
* Right handed
* Learned English prior to age 5
* Agrees to use an effective form of contraception throughout the study

For healthy controls:

* Medically healthy
* Right handed
* Has experienced a qualifying traumatic event
* Does not meet DSM-IV criteria for present or past PTSD
* Learned English prior to age 5
* Agrees to use an effective form of contraception throughout the study

Exclusion Criteria:

For people with PTSD:

* Meets DSM-IV criteria for panic disorder within 6 months prior to study entry
* Current suicide risk
* History of DSM-IV diagnosis of any the following conditions: schizophrenia, bipolar mood disorder, obsessive compulsive disorder (including trichotillomania), or eating disorder
* Meets DSM-IV criteria for substance use or dependence within the 6 months prior to study entry
* Any substance abuse within 2 weeks prior to study entry
* Score of greater than 22 on the 17-item Hamilton Rating Scale for Depression (HAM-D) with depressive symptoms secondary to PTSD
* Current participation in cognitive behavioral psychotherapy that is specifically designed to treat PTSD
* Concomitant psychoactive medications
* History of cerebrovascular accident (CVA) or any disorder that causes chronic neurological problems
* Medical illness with central nervous system (CNS) involvement or currently taking medication that affects the CNS
* Unstable general medical illness requiring intervention (e.g., HIV infection)
* Pregnant, breastfeeding, or plans to become pregnant
* Presence of internal metallic objects, such as heart pacemaker, shrapnel, bullets, surgical prostheses, surgical clips, or pins
* History of gastric bypass surgery

For healthy controls:

* Any history of generalized anxiety disorder or panic disorder
* Any history of psychotic disorder, bipolar disorder, or cyclothymia
* Any history of substance abuse or dependence within the 6 months prior to study entry
* Any substance use within 2 weeks prior to study entry
* Any other Axis I disorder within the year prior to study entry, including obsessive-compulsive disorder and trichotillomania
* Unstable general medical illness requiring intervention (e.g., HIV infection)
* Presence of internal metallic objects, such as heart pacemaker, shrapnel, bullets, surgical prostheses, surgical clips, or pins
* Concomitant psychoactive medications
* Patients with a history of cerebrovascular accident (CVA) or any disorder that causes chronic neurological problems
* Medical illness with central nervous system (CNS) involvement or currently taking medication that affects the CNS
* Cognitive impairment or severe Axis II disorder that will likely affect participation in the study
* Pregnant, breastfeeding, or plans to become pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2005-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marylene Cloitre, PhD, Principal Investigator — NYU
Locations (1):
- NYU Institute for Trauma & Resilience, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Behavioral Therapy: Participants will receive cognitive behavioral therapy
  Cognitive behavioral therapy (CBT): CBT consists of sixteen 1-hour sessions during a period of 12 weeks.
Period: Overall Study
Arm/Group | Sertraline | Control | Cognitive Behavioral Therapy
Started | 8 | 0 | 31
Completed | 5 | 0 | 19
Not Completed | 3 | 0 | 12
Not completed — Withdrawal by Subject | 3 | 0 | 12

BASELINE CHARACTERISTICS:
Population: Multiple efforts were made to locate the study data, but were unsuccessful (study was terminated, data was not saved). No study data are available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy | Total
Number analyzed (Participants) | 0 | 8 | 31 | 39
Age, Continuous [Mean (Full Range); unit: years] — Age assessed in years Population: Study was terminated due to poor enrollment. Data collected insufficient to conduct meaningful analyses.
Sex: Female, Male [Count of Participants; unit: Participants] — Gender specified by status of either being male or female. Population: Multiple efforts were made to locate the study data, but were unsuccessful (study was terminated, data was not saved). No study data are available.

OUTCOME MEASURES:

1. Primary Outcome: Salivary Cortisol Levels (Measured Before, During, and After the fMRI)
Description: Salivary cortisol levels (measured before, during, and after the fMRI)
Time Frame: Measured 3 days before and after treatment and 1 day during fMRI
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Fear Response (Measured During the fMRI)
Description: Fear response (measured during the fMRI) in response to positive fearful and neutral stimuli
Time Frame: Measured on 1 day during two MRIs
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Trauma History Inventory (THI)
Description: Assesses the full range of traumatic stressor over lifetime
Time Frame: Measured 30 minutes before and after treatment
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Clinician-Administered PTSD Scale for DSM-IV (CAPS)
Description: Assesses severity and frequency of PTSD symptoms and provides information for diagnosis
Time Frame: Measured 30 minutes before and after treatment
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Structured Clinical Interview for DSM-IV I and II (SCID I and II)
Description: Provides assessment of all anxiety and mood disorder diagnoses
Time Frame: Measured 1 hour before and after treatment
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Panic Disorder Severity Scale (PDSS)
Description: measure of frequency and severity of panic attacks
Time Frame: Measured 15 minutes before and after treatment
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Clinical Global Impressions Severity Scale
Description: Assesses functional status of individual
Time Frame: Measured weekly throughout the study
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Clinical Global Impressions Improvement Scale
Description: Assesses improvement in functioning
Time Frame: Measured weekly throughout the study
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Sociodemographic Questionnaire
Description: social and demographic characteristics of the individual
Time Frame: Measured at baseline
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Penn State Worry Questionnaire (PSWQ)
Description: assesses worry and rumination
Time Frame: Measured 10 minutes, before, during, and after treatment
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Post Traumatic Stress Disorder Symptom Scale-Self Report (PSS-SR)
Description: self-report measure of PTSD symptoms
Time Frame: Measured 10 times throughout study
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Brief Symptom Inventory (BSI)
Description: assesses a wide range of symptoms regarding the distress they cause
Time Frame: Measured 10 times throughout study
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: General Expectancy for Negative Mood Regulation (NMR)
Description: assesses ability to regulate mood states
Time Frame: Measured 3 times throughout study
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: State-Trait Anger Expression (STAXI)
Description: assess experience of anger as both a state and trait like phenomenon
Time Frame: Measured 10 times throughout study
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Toronto Alexithymia Scale (TAS)
Description: assesses difficulty in identifying and naming feelings
Time Frame: Measured 2 times throughout study
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: The State-Trait Anxiety Inventory (STAI)
Description: assesses types and severity of anxiety
Time Frame: Measured 10 times throughout study
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Beck Depression Inventory (BDI)
Description: assesses type and severity of depression
Time Frame: Measured 3 times throughout study
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

18. Secondary Outcome: The Inventory of Interpersonal Problems (IIP)
Description: assesses type and severity of interpersonal problems
Time Frame: Measured 2 times throughout study
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: The Social Adjustment Scale - Self Report (SAS-SR)
Description: assesses social adjustment
Time Frame: Measured 2 times throughout study
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: fMRI Safety Information Checklist
Description: review safety information related to fMRI procedure
Time Frame: Measured 2 times throughout study
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

21. Secondary Outcome: Medical History 12 Months (MH)
Description: assessment of medical problems in past 12 months
Time Frame: Measured throughout study
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

22. Secondary Outcome: Health Services Utilization Form-12 Months (HSUF)
Description: assessment of type and frequency of use of medical services
Time Frame: Measured throughout study
Population: as for baseline characteristics
Arm/Group | Control | Sertraline | Cognitive Behavioral Therapy
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 4 years
Description: 0 participants completed in control arm; therefore 0 participants at risk for adverse events
Arm/Group | Sertraline | Control | Cognitive Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0 | 0/12
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No